CLINICAL TRIAL: NCT00207220
Title: Ventricular-Vascular Coupling in Patients With Heart Failure and Preserved Ejection Fraction
Brief Title: Ventricular-Vascular Coupling in Heart Failure
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Other Study IDs: 2003P-001769
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure; preserved ejection fraction; vascular stiffness
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3: subjects with heart failure and normal ejection fraction non-diabetic hypertensive controls hypertensive diabetic controls normotensive controls
  Interventions: Procedure: arterial tonometry; Procedure: echocardiography

INTERVENTIONS:
Procedure: arterial tonometry — used to determine peripheral arterial vascular tone by measuring blood pressure waveforms via a probe attached to the finger.
  Other Names: PAT
Procedure: echocardiography — ultrasound test using sound waves to create a moving picture of the heart
  Other Names: cardiac echo

SUMMARY:
This study will test the hypothesis that increases in ventricular-vascular stiffness can be demonstrated by arterial tonometry and echocardiography in subjects with heart failure with preserved ejection fraction (HF-nlEF)(i.e. normal left ventricular function.) We will also track changes in pulsatile hemodynamics over time in subjects hospitalized with HF-nlEF.

DETAILED DESCRIPTION:
The pathophysiologic mechanisms responsible for the development of heart failure in people with preserved ejection fraction (i.e. normal left ventricular function) remain poorly understood. One possible mechanism may be the contribution of increased arterial stiffness to changes in pulsatile hemodynamic load during ventricular systole, implicating abnormal ventricular-vascular interactions throughout the cardiac cycle in the pathogenesis of heart failure with normal ejection fraction.

To investigate changes in ventricular-vascular stiffness in subjects with heart failure and normal left ventricular function, comparisons will be made between 3 distinct sub-populations:

* subjects with heart failure and normal ejection fraction
* non-diabetic hypertensive controls
* normotensive controls

ELIGIBILITY:
Inclusion Criteria:

Subjects with heart failure and preserved ejection fraction

* clinical signs of heart failure
* serum brain natriuretic peptide (BNP) >100pg/mL
* NYHA functional class II-IV
* left ventricular ejection fraction(LVEF) >=50% measured by echocardiography
* Non-diabetic subjects with hypertension
* treated or untreated essential hypertension
* LVEF >=50% measured by echocardiography

Diabetic subjects with hypertension

* Type 2 diabetes
* treated or untreated essential hypertension
* LVEF >=50% measured by echocardiography

Normotensive control subjects

* normal blood pressure (i.e. < 140/90 mmHg)
* LVEF >=50% measured by echocardiography

Exclusion Criteria:

Subjects with heart failure and preserved ejection fraction

* atrial fibrillation
* symptoms of angina or a myocardial infarction (MI) within 6 months
* known significant coronary artery disease (CAD) (stenosis > 70%)
* significant valvular heart disease
* restrictive/constrictive heart disease
* inability to lie flat for procedure (estimated duration 1 hour)

Non-diabetic subjects with hypertension

* atrial fibrillation
* symptoms of angina or a myocardial infarction (MI) within 6 months
* known significant coronary artery disease (CAD) (stenosis > 70%)
* significant valvular heart disease
* restrictive/constrictive heart disease
* inability to lie flat for procedure (estimated duration 1 hour)
* prior history of heart failure or unexplained dyspnea

Diabetic subjects with hypertension

* atrial fibrillation
* symptoms of angina or a myocardial infarction (MI) within 6 months
* known significant coronary artery disease (CAD) (stenosis > 70%)
* significant valvular heart disease
* restrictive/constrictive heart disease
* inability to lie flat for procedure (estimated duration 1 hour)
* prior history of heart failure or unexplained dyspnea

Normotensive control subjects

* prior history of structural heart disease or ventricular hypertrophy
* treatment with HMG-Co(A)reductase inhibitors (statins)
* anti-hypertensive medications
* cigarette smoking
* cocaine use
* excessive alcohol intake

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with heart failure and preserved left ventricular function
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2004-01; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Creager, M.D., Principal Investigator — Brigham and Women's Hospital; Akshay S. Desai, M.D., Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States